CLINICAL TRIAL: NCT06711328
Title: Effect of New Oropharyngeal Airway on Incidence of Hypoxia During Painless Gastroenteroscopy in Elderly Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jianbo Wu (Other)
Responsible Party: Sponsor-Investigator, Jianbo Wu, chief physician, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: YXLL-KY-2024(083)
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Airway Management; Elderly Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Using a new oropharyngeal airway set (Experimental): Study participants entered the examination room to establish intravenous access, using 2% lidocaine gel 5ml containing mouth cavity and pharynx.Heart rate (HR), pulse oxygen saturation (SpO2), end-expiratory carbon dioxide, ECG monitoring, and non-invasive blood pressure (measured every 2.5 minutes) were routinely monitored before anesthesia induction.Study participants were asked to lie on their left side.In this study, the relevant staff of the undergraduate department participating in this clinical trial planned to implement simple randomization using SAS: The group using the new oropharyngeal airway (trial group) : Oxygen was continuously supplied through a catheter partially connected to the endoscopic mouth before induction of anesthesia until the end of gastroenteroscopy
  Interventions: Device: New oropharyngeal airway
- The conventional endoscopic bite group (No Intervention): Study participants entered the examination room to establish intravenous access, using 2% lidocaine gel 5ml containing mouth cavity and pharynx.Heart rate (HR), pulse oxygen saturation (SpO2), end-expiratory carbon dioxide, ECG monitoring, and non-invasive blood pressure (measured every 2.5 minutes) were routinely monitored before anesthesia induction.Study participants were asked to lie on their left side.In this study, the relevant staff of the undergraduate department participating in this clinical trial planned to implement simple randomization using SAS:In the conventional endoscopic bite group (control group), oxygen was continuously supplied through a common nasal catheter before induction of anesthesia until the end of gastroenteroscopy.

INTERVENTIONS:
Device: New oropharyngeal airway — This product is produced and sold by Shanghai Elifu Medical Technology Co., LTD., and has been officially put into clinical use in March 2023.The product is named oropharyngeal airway for disposable endoscope, which is composed of nasal plug, bite, oropharyngeal channel, oxygen supply tube, lanyard and optional accessories carbon dioxide gas catheter and carbon dioxide collection tube.The model used in this study is JK (Oropharyngeal airway for endoscope with end-expiratory carbon dioxide Collection) with L/M/S three specifications, which is used to prevent airway obstruction caused by backward tongue fall during endoscopic surgery/examination, establish oropharyngeal airway for patients, and provide nasal oxygen at the same time
  Arms: Using a new oropharyngeal airway set

SUMMARY:
With the aging of Chinese population, the early screening of gastrointestinal diseases and the promotion and implementation of comfortable medical treatment, more and more elderly patients choose painless gastroenteroscopy for diagnosis and treatment.However, the incidence of anesthesia-related adverse reactions and complications is high in elderly patients.Hypoxemia caused by anesthetic-induced respiratory depression and airway obstruction is a serious complication in painless gastroenteroscopy.Severe hypoxemia not only requires emergency airway intervention, such as mask ventilation or even tracheal intubation, but also leads to the interruption of endoscopic diagnosis and treatment.Advanced age was an independent risk factor for hypoxemia during painless gastroenteroscopy,This study observed the effect of a new type of oropharyngeal ventilation in improving the elderly painless gastroenteroscopy anesthesia hypoxemia and reducing intraoperative airway intervention, so as to evaluate the safety and effectiveness of a new type of nasopharyngeal ventilation in the elderly painless gastrointestinal diagnosis and treatment, and provide clinical reference.

DETAILED DESCRIPTION:
The oropharyngeal airway is an important airway auxiliary device for short-term airway management during the perianesthetic period, which can provide patients with an unobstructed airway during autonomous ventilation .The oropharyngeal vent has been proven to be successfully used in infants, the elderly and MRI, and can be used in short outpatient surgery instead of laryngeal mask .The oropharyngeal airway has a low incidence of pharyngeal trauma and laryngeal pain immediately after surgery, requiring a shorter exposure time of inhaled anesthetic and a lower concentration of propofol to successfully place it .During the operation to preserve spontaneous breathing, the oropharyngeal airway is introduced as a ventilation device .The new oropharyngeal airway can accept the implantation of gastroscopy and provide oxygen to patients without affecting the operation at the same time. In order to explore whether the new oropharyngeal airway can provide better oxygen to patients undergoing painless gastroenteroscopy and reduce the incidence of hypoxia during the operation, we have drafted this study and explored the safety of the new oropharyngeal airway in painless gastroenteroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Age 65-80 years old
* written informed consent of patient or family member
* painless stomach + colonoscopy
* ASA grade I-II

Exclusion Criteria:

* Patients with clotting disorders or a tendency to oropharyngeal bleeding, mucosal damage or space occupation, difficulty in placing oropharyngeal airway, etc., who could not perform oropharyngeal airway ventilation;
* Upper respiratory tract infections such as mouth, nose or throat;
* Fever (core body temperature ≥37.5℃);
* a confirmed diagnosis of pregnancy or breastfeeding;
* Allergic to sedatives such as propofol or equipment such as tape;
* Emergency surgery;
* Multiple trauma;
* SpO2 < 95% before operation;
* A history of drug and/or alcohol abuse within 2 years prior to the start of the screening period;(Drinking more than three times standard alcoholic beverages per day, equivalent to about 10g of alcohol or equivalent to 50g of Chinese liquor);
* Patients with previous psychiatric and neurological diseases, such as depression, severe central nervous depression, Parkinson's disease, basal ganglia disease, schizophrenia, epilepsy, Alzheimer's disease, myasthenia gravis;
* Currently participating in other clinical trials;
* Patients who are deemed unfit by the investigator to participate in the trial;
* Patients with a history of smoking should not participate in this study.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of hypoxia | 1 minute after anesthesia induction
  The incidence of hypoxia (75% ≤ SpO2 < 90%, ≤ 60s)

SECONDARY OUTCOMES:
The incidence of severe hypoxia | 1 minute after anesthesia induction
  The incidence of severe hypoxia (SpO2 < 75% or 75% ≤SpO2 < 90%, ≥60s)
The incidence of requiring airway intervention | 1 minute after anesthesia induction
  Tracheal intubation and noninvasive ventilation are required
Cyclic fluctuation | 1 minute after anesthesia induction
  Severe bradycardia (< 50 beats/min), MAP fluctuation greater than 30% of the baseline value or MAP < 60 mmHg
The satisfaction of endoscopists was recorded | Within 30 minutes after anesthesia awakening
  Patient satisfaction scales usually use a 0-10 scale, where 0 is very dissatisfied and 10
Recorded adverse events | 1 minute after anesthesia induction
  The incidence of choking, laryngeal spasm and reflux aspiration were observed.Apnea or slow breathing episodes (defined as respiratory rate ≤6 beats/min);Bradycardia is defined as a heart rate ≤50 beats/min.Serious adverse events such as tracheal intubation, non-invasive ventilation, use of vasopressors, and hospitalization are required.

CONTACTS AND LOCATIONS:
Overall Officials: Jianbo Wu, Doctoral, Study Director — Department director

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] You Q, Meng Y, Liu X, Sun C, Wu J. Clinical efficacy of COMBO endoscopy of oropharyngeal airways in elderly patients undergoing painless gastroenteroscopy under anaesthesia: a randomized controlled trial protocol. BMC Anesthesiol. 2025 Sep 26;25(1):453. doi: 10.1186/s12871-025-03311-8. PMID 41013276